CLINICAL TRIAL: NCT00197080
Title: A 12-Week, Double-Blind, Placebo Controlled, Parallel Group Study to Assess the Efficacy and Safety of Ropinirole XR (Extended Release) in Patients With Restless Legs Syndrome
Brief Title: Ropinirole XR (Extended Release) In Patients With Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101468/205
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole Extended Release (XR)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ropinirole XR in the treatment of adults with Restless Legs Syndrome (RLS).

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with RLS using the International RLS Study Group Diagnostic Criteria with a total score of 15 or greater on the International RLS Rating Scale.
* Have evening and nighttime symptoms of RLS, significant sleep impairment due to RLS symptoms, and symptoms requiring treatment prior to bedtime, but no earlier than 5:00PM.

Exclusion criteria:

* Have secondary RLS.
* Have any medical conditions that may impact efficacy assessments or that may present a safety concern.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline in the International RLS Study Group Rating Scale total score at Week 12. | 12 Weeks

SECONDARY OUTCOMES:
Assess safety, tolerability, and patient-reported outcomes, including changes in the Clinical Global Impression Scale Scores and changes in the Medical Outcomes Study Sleep Scale at Week 12. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- United States (58):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Dawsonville, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Northbrook, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Canada (9):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register